CLINICAL TRIAL: NCT07207031
Title: Acute Kidney Injury - Epidemiology in Intensive Care Unit Patients 2
Brief Title: Acute Kidney Injury - Epidemiology in Intensive Care Unit Patients 2: an International Multicenter Cohort Study
Acronym: AKI-EPI2
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Tirol Kiniken GmbH (Other); Austin Hospital, Melbourne Australia (Other); Hospices Civils de Lyon (Other); Royal Surrey County Hospital NHS Foundation Trust (Other); University of Alberta (Other); Universitätsklinkum Münster - Medizinische Klinik und Poliklinik B (Other); St. Bartholomew's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0185
Record Dates: First submitted 2024-12-04; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Kidney Injury, Acute; Intensive Care Unit ICU
Keywords: Acute Kidney Injury; Intensive Care Unit; Epidemiology; major adverse kidney events
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive Care Unit patients: adult patients admitted to the intensive care unit

SUMMARY:
The goal of this observational study is to learn the epidemiology and outcomes of acute kidney injury in critically ill adult patients admited to the intensive care unit (ICU). The main questions it aims to answer are:To provide a contemporary update on the epidemiology (rates, severity, duration, and etiology) of acute kidney injury and associated outcomes in critically ill patients.

The co-primary outcomes are:

* occurrence rate of acute kidney injury within 7 days of ICU admission
* maximum severity of acute kidney injury within 7 days of ICU admission.

Secondary outcomes:

* Proportion of acute kidney injury in patients with and without known baseline serum creatinine
* Duration of acute kidney injury episodes (within first week of ICU admission)
* Proportion of episodes with rapid reversal (duration <48h) versus persistent acute kidney injury (duration ≥48h)
* Incidence of acute kidney disease at ICU discharge and hospital discharge, truncated at 90-d
* Use of Renal Replacement Therapy within 7 days of ICU admission
* Type and specifics of applied Renal Replacement Therapy (indications, timing, modality, method duration, anticoagulation, discontinuation)
* ICU lenght of stay (ICU LOS), Hospital lenght of stay (Hospital LOS)
* ICU readmission up to day 90
* Hospital readmission up to day 90
* Serum creatinine level at ICU and hospital discharge (truncated at day 90)
* RRT dependence at hospital discharge (any RRT applied within 72 hours of discharge)
* Mortality at hospital discharge (truncated at 90-d)
* Magnitude of acute kidney injury: area under the curve of acute kidney injury severity over time
* Incidence of acute kidney injury and maximum acute kidney injury severity stage defined by serum creatinine and/or urine output criteria only, within 7 days of ICU admission.

Additional endpoints for patients included in the "long term outcomes substudy":

* Serum creatinine level at day 90, and 1 y
* Renal Replacement Therapy dependence at day 90, and 1y
* Mortality at hospital discharge at day 90, and 1y
* Survival analysis up to day 90 and 1 y
* Health-related quality of life at day 90 and 1y
* Major Adverse Kidney Events (MAKE): a composite endpoint of death, use of Renal Replacement Therapy and decreased kidney function at day 90, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 y
* Admitted to a participating ICU.
* Admitted to the ICU for more than 24-h, or anticipated length of stay in the ICU for 24-h or more.
* Informed Consent according to local ethical committee

Exclusion Criteria:

* End Stage Kidney Disease treated with maintenance renal replacement therapy
* Readmission to the ICU during same hospitalization episode
* Missing acute kidney injury defining data (no measured serum creatinine and <6 hours of documented urinary output)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 10642 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
occurrence rate of acute kidney injury | within 7 days of ICU admission
  occurrence rate of acute kidney injury in adult patients admitted to the ICU and defined by the Kidney Disease: Improving Global Outcomes defintion
maximum severity of acute kidney injury | within 7 days of ICU admission.
  maximum severity of acute kidney injury defined by the Kidney Disease: Improving Global Outcomes classification

SECONDARY OUTCOMES:
Proportion of acute kidney injury in patients with and without known baseline serum creatinine | within 7 days of ICU admission.
  acute kidney injury as defined by the Kidney Disease: Improving Global Outcomes definition in patients with known baseline serum creatinine and in those without known baseline serum creatinine
Duration of acute kidney injury episodes | within 7 days of ICU admission.
  acute kidney injury defined by the Kidney Disease: Improving Global Outcomes definition, and duration measured in days
Proportion of episodes with rapid reversal (duration <48h) and persistent acute kidney injury(duration ≥48h) | within 7 days of ICU admission.
  acute kidney injury defined by the Kidney Disease: Improving Global Outcomes definition
Incidence of acute kidney disease | at ICU discharge and at hospital discharge, or at 90-days in case hospital admission is longer than 90 days.
  acute kidney disease as defined by the Kidney Disease: Improving Global Outcomes definition
Use of renal replacement therapy within 7 days of ICU admission | within 7 days of ICU admission.
Type and specifics of applied renal replacement therapy | within 7 days of ICU admission.
  indications, timing, modality, method duration, anticoagulation, discontinuation
Length of stay | hospital stay
  Length of stay in the ICU, post ICU in the hospital, and total length of stay in the hospital , measured in days
ICU readmission up to day 90 | within 90 days of ICU admission
Hospital readmission up to day 90 | within 90 days of ICU admission
Serum creatinine level at ICU and hospital discharge (truncated at day 90) | at discharge of the ICU and of the hospital, or day 90 after ICU admission if hospital stay is longer than 90 days after ICU admission
Renal Replacement Therapy dependence at hospital discharge | hospital discharge
  Renal Replacement Therapy dependence is defined as the use of renal replacement therapy within 72-hours before hospital discharge
Mortality | at hospital discharge or at day 90 after ICU admission if hospital stay is longer than 90 days after ICU admission
Magnitude of acute kidney injury | within 7 days of ICU admission.
  Magnitude of acute kidney injury: defined as the area under the curve of acute kidney injury severity over time
Incidence of acute kidney injury and maximum acute kidney injury severity stage defined by serum creatinine criteria only and urine output criteria only | within 7 days of ICU admission.
  acute kidney injury is defined and classified by the Kidney Disease: Improving Global Outcomes definition

OTHER OUTCOMES:
Serum creatinine level at day 90, and at1 year | at 90 days after ICU admission and at 1 year after ICU admission
Renal Replacement Therapy dependence | at 90 days after ICU admission and at 1 year after ICU admission
Mortality | at 90 days after ICU admission and at 1 year after ICU admission
Survival | at 90 days after ICU admission and at 1 year after ICU admission
Health-related quality of life | at 90 days after ICU admission and at 1 year after ICU admission
  Measured with the EuroQol-5D-5L instrument
Major Adverse Kidney Events (MAKE): | at 90 days after ICU admission and at 1 year after ICU admission
  Major Adverse Kidney Events (MAKE): a composite endpoint of death, use of RRT and decreased kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, MD, PhD, Principal Investigator — University Hospital, Ghent; Antoine Schneider, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vandois (CHUV)
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- See also: Related Info — https://www.ualberta.ca/en/critical-care/research/aki-epi-2/index.html